CLINICAL TRIAL: NCT02671812
Title: Longterm Outcome After Dental Implant Treatment
Brief Title: Outcome After Dental Implant Treatment
Status: Completed | Type: Observational
Sponsor: Folktandvården Stockholms län AB (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Leif Jansson, DDS PhD-student, Folktandvården Stockholms län AB
Other Study IDs: OF13122003
Record Dates: First submitted 2016-01-30; First posted 2016-02-02 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2019-02

CONDITIONS: PROMs; Peri-implantitis; Mucositis; Periodontitis
Keywords: dental implant; patient satisfaction; treatment outcome; cytokine profile; risk factor; risk predictor
MeSH Terms: conditions — Peri-Implantitis; Mucositis; Periodontitis; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and gingival fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The general aim of this project is to investigate the long-term treatment outcome after implant therapy. The patients' satisfaction with implant treatment will be studied and correlated to biological and technical problems. The survival rates of implants at patient level and the degree of bone loss of remaining teeth and implants will be calculated. The levels of cytokines and bone loss markers in peri-implantitis sites and periodontal defects and at healthy sites will be analyzed in order to study the correlation between cytokine and bone loss marker levels, and clinical conditions. Independent variables which could be regarded as significant risk factors or risk predictors on the incidence of peri-implantitis are aimed to be identified

DETAILED DESCRIPTION:
* A questionnaire study will investigate patient satisfaction 8-14 years after dental implant therapy to study if complications influence the degree of satisfaction/quality of life. The questionnaire will be sent to 587 patients treated at The Specialist Clinic Skanstull.
* A clinical examination of a minimum 150 patients who answered the questionnaire will be performed:
* to study the incidence of biological and technical complications on dental implants after a minimum of 10 year of function.
* to study the survival rates of implants at patient level and the degree of bone loss of remaining teeth and implants. In addition, the correlation between bone loss of remaining teeth and bone loss of implants will be studied.
* samples taken from the gingival crevicular fluid to investigate the profile of cytokines and bone resorption markers as well as to study the intra-individual correlation of cytokines and bone markers in gingival crevicular fluid from sites with peri-implantitis and periodontal defects in individuals with dental implants.
* in addition, the salivary cytokine and bone resorption markers will be analyzed in order to identify disease-specific biomarkers as well as to study the correlation between the cytokine/bone resorption markers in saliva and in gingival/peri-implant crevicular fluid.
* To identify significant risk factors or risk predictors on the incidence of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

- Treated at the Specialist Clinic Skanstull, Stockholm, Sweden with dental implants between the years of 1999-2005

Exclusion Criteria:

- Deceased before or during the study period

Ages: 20 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with dental implants at the Specialist Clinic Skanstull, Stockholm, Sweden, between 1999-2005
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2014-11-27 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Patients satisfaction after dental implant treatment | 10 years after implant treatment
  Questionnaire and clinical examination

SECONDARY OUTCOMES:
Complications prevalence | 10 years after implant treatment
  Self reported and registered in patients journal and detected at the clinical examination
Profile of inflamatory markers | 10 years after implant treatment
  Samples of saliva and gingival fluid from healthy and disease sites at both tooth and dental implants will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Sällberg Chen, Assc. Prof, Study Director — Karolinska Institutet Odontologen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Result] Pjetursson BE, Karoussis I, Burgin W, Bragger U, Lang NP. Patients' satisfaction following implant therapy. A 10-year prospective cohort study. Clin Oral Implants Res. 2005 Apr;16(2):185-93. doi: 10.1111/j.1600-0501.2004.01094.x. PMID 15777328
- [Result] Derks J, Hakansson J, Wennstrom JL, Klinge B, Berglundh T. Patient-reported outcomes of dental implant therapy in a large randomly selected sample. Clin Oral Implants Res. 2015 May;26(5):586-91. doi: 10.1111/clr.12464. Epub 2014 Aug 14. PMID 25123298
- [Result] Heitz-Mayfield LJ. Peri-implant diseases: diagnosis and risk indicators. J Clin Periodontol. 2008 Sep;35(8 Suppl):292-304. doi: 10.1111/j.1600-051X.2008.01275.x. PMID 18724857
- [Result] Roccuzzo M, Bonino F, Aglietta M, Dalmasso P. Ten-year results of a three arms prospective cohort study on implants in periodontally compromised patients. Part 2: clinical results. Clin Oral Implants Res. 2012 Apr;23(4):389-95. doi: 10.1111/j.1600-0501.2011.02309.x. Epub 2011 Sep 28. PMID 22092445
- [Result] Andreiotelli M, Koutayas SO, Madianos PN, Strub JR. Relationship between interleukin-1 genotype and peri-implantitis: a literature review. Quintessence Int. 2008 Apr;39(4):289-98. PMID 19081897
- [Result] Sharma CG, Pradeep AR. Plasma and crevicular fluid osteopontin levels in periodontal health and disease. J Periodontal Res. 2007 Oct;42(5):450-5. doi: 10.1111/j.1600-0765.2007.00968.x. PMID 17760823